CLINICAL TRIAL: NCT01949909
Title: Safety And Immunogenicity Of Novel Candidate Blood-Stage Malaria Vaccine P27A With Alhydrogel® Or GLA-SE As Adjuvant: A Staggered, Antigen And Adjuvant Dose-Finding, Randomized, Multi-Centre Phase Ia/Ib Trial
Brief Title: Safety And Immunogenicity Of Novel Candidate Blood-Stage Malaria Vaccine P27A : Phase Ia/Ib
Acronym: P27A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: European Vaccine Initiative (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Principal Investigator, François Spertini, Dr, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P27A_1_13
Record Dates: First submitted 2013-08-29; First posted 2013-09-25 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Malaria
Keywords: plasmodium falciparum; long synthetic peptide; antibody; T cell; cytokine; vaccine; safety; phase 1
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Alhydrogel CH-Alum50 (Experimental): intramuscular administration to Swiss volunteers of Alhydrogel and P27A antigen (50 microg)
  Interventions: Biological: CH-Alum50
- CH-GLA2.5/50 (Experimental): intramuscular administration to Swiss volunteers of GLA-SE (2.5microg) together with the P27A antigen (50 microg)
  Interventions: Biological: CH-GLA2.5/50
- Control rabies vaccine Verorub TM TZ Ver (Placebo Comparator): intramuscular administration of Rabies vaccine Verorub TM to in Phase IIb only to 8 Tanzanian volunteers in three injections
  Interventions: Biological: TZ Ver
- Alhydrogel TZ Alum 50 (Experimental): intramuscular administration to Tanzanian volunteers of Alhydrogel and P27A antigen (50 microg)
  Interventions: Biological: TZ Alum 50
- GLA-SE TZ GLA 2.5/10 (Experimental): intramuscular administration to Tanzanian volunteers of GLA-SE (2.5 microg ) together with the P27A antigen (10 microg)
  Interventions: Biological: TZ GLA 2.5/10
- GLA-SE TZ GLA5/50 (Experimental): intramuscular administration to Tanzanian volunteers of GLA-SE (5 microg) together with the P27A antigen (50 microg)
  Interventions: Biological: TZ GLA5/50
- GLA-SE TZ GLA2.5/50 (Experimental): intramuscular administration to Tanzanian volunteers of GLA-SE (2.5microg) together with the P27A antigen (50 microg)
  Interventions: Biological: TZ GLA2.5/50

INTERVENTIONS:
Biological: CH-Alum50 — intramuscular administration to Swiss volunteers of Alhydrogel and P27A antigen (50 microg)
  Arms: Alhydrogel CH-Alum50
Biological: CH-GLA2.5/50 — intramuscular administration to Swiss volunteers of GLA-SE (2.5microg) together with the P27A antigen (50 microg)
  Arms: CH-GLA2.5/50
Biological: TZ Ver — intramuscular administration of Rabies vaccine Verorub TM to in Phase IIb only to 8 Tanzanian volunteers in three injections
  Arms: Control rabies vaccine Verorub TM TZ Ver
Biological: TZ Alum 50 — intramuscular administration to Tanzanian volunteers of Alhydrogel and P27A antigen (50 microg)
  Arms: Alhydrogel TZ Alum 50
Biological: TZ GLA 2.5/10 — intramuscular administration to Tanzanian volunteers of GLA-SE (2.5 microg ) together with the P27A antigen (10 microg)
  Arms: GLA-SE TZ GLA 2.5/10
Biological: TZ GLA5/50 — intramuscular administration to Tanzanian volunteers of GLA-SE (5 microg) together with the P27A antigen (50 microg)
  Arms: GLA-SE TZ GLA5/50
Biological: TZ GLA2.5/50 — intramuscular administration to Tanzanian volunteers of GLA-SE (2.5microg) together with the P27A antigen (50 microg)
  Arms: GLA-SE TZ GLA2.5/50

SUMMARY:
P27A study is designed as a randomized phase Ia/Ib trial to evaluate the safety and immunogenicity of the blood stage candidate vaccine P27A against P. falciparum - P27A antigen and associated adjuvant (Alhydrogel or GLA-SE) - in malaria non exposed European volunteers(Switzerland; phase Ia) and malaria exposed African volunteers (Tanzania; phase Ib).

ELIGIBILITY:
Inclusion Criteria:

* Phase Ia Inclusion criteria:

  1. Healthy volunteers aged 18-45 years
  2. General good health based on history and clinical examination
  3. Written informed consent obtained before any study procedure
  4. Female volunteers practicing contraception before and up to 13 weeks after the last immunisation
  5. Available to participate in follow-up for the duration of study (34 weeks)
  6. Reachable by phone during the whole study period
* Phase Ib inclusion criteria

  1. Healthy male volunteers aged 18-45 years
  2. General good health based on history and clinical examination
  3. Written informed consent obtained before any study procedure
  4. Available to participate in follow-up for the duration of study (34 weeks)
  5. Reachable by phone during the whole study period
  6. Having always lived in an area of low malaria transmission

Exclusion Criteria:

* Phase Ia Exclusion criteria:

  1. Positive pregnancy test for females
  2. Actively breast feeding females
  3. Previous participation in any malaria vaccine trial
  4. Symptoms, physical signs or laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the trial results or compromise the health of the volunteers
  5. Any clinically significant laboratory abnormalities on screened blood samples beyond the normal range, as defined at the clinical trial site
  6. Enrolment in any other clinical trial during the whole trial period
  7. Intake of chronic medication, especially immunosuppressive agents (steroids, immunomodulating or immunosuppressive drugs) during the 13 weeks preceding the screening visit or during the trial period except topical and inhaled steroids
  8. Volunteers unable to be closely followed for social, geographic or psychological reasons
  9. Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the study
  10. Known hypersensitivity to any of the vaccine components (adjuvant or peptide)
  11. Vaccination or infusion of gammaglobulin from 4 weeks prior to the first vaccination and up to 6 weeks after the third vaccination
  12. Any history of malaria
  13. History of living in a malaria endemic area for more than five (5) years OR living in a malaria endemic area in early childhood. For practical purposes, all regions for which malaria chemoprophylaxis is advised by travel clinic are considered malaria endemic (cf. www.safetravel.ch).
  14. Known exposure to malaria in the previous six (6) months, defined as a visit to a malaria endemic region
  15. P27A ELISA positive OR parasite ELISA antibody positive AND Known exposure to malaria in a malaria endemic area
  16. P27A ELISA positive AND parasite ELISA antibody positive (with or without history of stay in a malaria endemic area)
  17. Intention to travel to malaria endemic countries during the study period
  18. Positive HIV, HBV or HCV tests
* Phase Ib exclusion criteria

  1. Previously participated in any malaria vaccine trial
  2. Symptoms, physical signs or laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the trial results or compromise the health of the volunteers
  3. Any clinically significant laboratory abnormalities on screened blood samples beyond the normal range, as defined at the clinical trial site
  4. Enrolment in any other clinical trial during the whole trial period
  5. Intake of chronic medication, especially immunosuppressive agents (steroids, immunomodulating or immunosuppressive drugs) during the thirteen weeks preceding the screening visit or during the trial period except topical and inhaled steroids
  6. Volunteers unable to be closely followed for social, geographic or psychological reasons
  7. Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the study
  8. Known hypersensitivity to any of the vaccine components (adjuvant or peptide) or to any of the control vaccine components
  9. Vaccination OR infusion of gammaglobulins from four (4) weeks prior to the first vaccination and up to six (6) weeks after the third vaccination
  10. Previous vaccination with the control vaccine
  11. Positive HIV, HCV test or HBVsAg positive
  12. Malaria parasite positivity by microscopy and/or RDT
  13. Having had a history of confirmed malaria episode in the last five year

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of P27A with Alhydrogel or GLA-SE as adjuvant, in healthy European adults not previously exposed to the parasite Plasmodium falciparum and in healthy African adults previously exposed to the parasite | 15 months
  The safety profile will be assessed on the basis of immediate local and systemic reactogenicity measured from Day 0 to Day 28 after each vaccination

SECONDARY OUTCOMES:
Assessment of the humoral immune response to the vaccine antigen | 15 months
  The humoral response to the vaccine antigen will be assessed in all volunteers by ELISA to measure the level of total antigen specific IgG.
Assessment of the cellular immune response to the vaccine antigen | 15 months
  The cellular immune response will be assessed in all volunteers by measuring the T cell proliferation and cytokine production following in vitro stimulation with the vaccine antigen (by Luminex on cell culture supernatant after in vitro stimulation of PBMC for 6 days with the P27A peptide). Proliferation of carboxyfluorescein diacetate succinimidyl ester (CFSE) loaded CD3+ CD4+ and CD3+CD8+ T cells will be assayed by using polychromatic flow cytometry.

OTHER OUTCOMES:
Exploratory outcome measure: humoral response | 15 months
  The humoral immune response quality will be assessed by measuring P27A specific antibodies IgG1, IgG2, IgG3, IgG4 subclasses by ELISA on samples obtained in all volunteers at day 0, week 8, week 12, week 26 and week 34.
Exploratory outcome measure: cytokine production (ICS) | 15 months
  The cellular immune response quality in all volunteers will be assessed by intracellular cytokine staining (ICS) for cytokines IL-2, TNF α, IFN γ and IL-10 in proliferating Carboxyfluorescein diacetate succinimidyl ester (CFSE) loaded CD3, CD4, and CD8 cells at day 0 and week 12 and 26.
Exploratory outcome measure : antibody dependent cell cytotoxicity (ADCI) | 15 months
  The functional humoral immune response will by ADCI in the GLA-SE and the Alhydrogel® group with the highest response, at day 0 and at an optimal time-point post vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: François Spertini, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV); Salim Abdulla, MD, Principal Investigator — Bagamoyo Research and Training Center
Locations (2):
- CHUV CRC, Lausanne, Switzerland
- Bagamoyo Clinical Trial Unit (BCTU), Bagamoyo, Tanzania

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Steiner-Monard V, Kamaka K, Karoui O, Roethlisberger S, Audran R, Daubenberger C, Fayet-Mello A, Erdmann-Voisin A, Felger I, Geiger K, Govender L, Houard S, Huber E, Mayor C, Mkindi C, Portevin D, Rusch S, Schmidlin S, Tiendrebeogo RW, Theisen M, Thierry AC, Vallotton L, Corradin G, Leroy O, Abdulla S, Shekalaghe S, Genton B, Spertini F, Jongo SA. The Candidate Blood-stage Malaria Vaccine P27A Induces a Robust Humoral Response in a Fast Track to the Field Phase 1 Trial in Exposed and Nonexposed Volunteers. Clin Infect Dis. 2019 Jan 18;68(3):466-474. doi: 10.1093/cid/ciy514. PMID 29945169
- See also: European Vaccine Initiative — http://www.euvaccine.eu